CLINICAL TRIAL: NCT01557465
Title: Study of Mechanical Alternans for Prediction of Ventricular Tachyarrhythmias
Brief Title: Mechanical Alternans Study
Acronym: MAS
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Larisa Tereshchenko, Instructor of Medicine, Johns Hopkins University
Other Study IDs: NA_00032758
Record Dates: First submitted 2012-03-16; First posted 2012-03-19 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Ischemic Cardiomyopathy; Nonischemic Cardiomyopathy; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether mechanical alternans (alternating strong and weak heart beats with a constant beat-to-beat interval), can be used to predict malignant ventricular arrhythmias, requiring defibrillation or appropriate ICD therapies, and to predict progression of heart failure and death.

ELIGIBILITY:
Inclusion Criteria:

* structural heart disease
* ischemic or non-ischemic cardiomyopathy

Exclusion Criteria:

* pregnancy
* age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with structural heart disease, ischemic or non-ischemic cardiomyopahty
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2009-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
sudden arrhythmic death | 5 years
  appropriate ICD therapy due to fast ventricular tachycardia or ventricular fibrillation, or sudden cardiac death

SECONDARY OUTCOMES:
cardiovascular mortality | 5 years
all-cause death | 5 years
appropriate ICD therapies | 5 years
  either ICD shock or antitachycardia pacing due to ventricular arrhythmia
composite heart failure endpoint | 5 years
  pump-failure death, or heart transplantation, or heart failure hospitalization, whichever came first

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Result] Kim R, Cingolani O, Wittstein I, McLean R, Han L, Cheng K, Robinson E, Brinker J, Schulman SS, Berger RD, Henrikson CA, Tereshchenko LG. Mechanical alternans is associated with mortality in acute hospitalized heart failure: prospective mechanical alternans study (MAS). Circ Arrhythm Electrophysiol. 2014 Apr;7(2):259-66. doi: 10.1161/CIRCEP.113.000958. Epub 2014 Mar 1. PMID 24585716